CLINICAL TRIAL: NCT04214509
Title: LIPAD - LRRK2 International Parkinson's Disease Study: an International, Multicenter, Epidemiological Observational Study
Brief Title: LIPAD - LRRK2 International Parkinson's Disease Study
Acronym: LIPAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Luebeck (Other)
Collaborators: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Principal Investigator, Meike Kasten, Prof., University of Luebeck
Other Study IDs: LIPAD
Record Dates: First submitted 2019-12-24; First posted 2020-01-02 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Parkinson's Disease and Parkinsonism
Keywords: genetic Parkinson's disease; LRRK2
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and urine samples will be biochemically analysed to determine factors leading to incomplete penetrance in LRRK2 positive carriers and biomarkers of Parkinson's disease.
  In blood samples DNA and DNA methylation, RNA and proteins will be analysed. Urine samples will be analysed using NGS-based sequencing of the mitochondrial genome and search for mitochondrial DNA deletions.
  Dust will be analysed toxicologically.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- PD + LRRK2: Patients with LRRK2-associated Parkinson's syndrome
- no PD + LRRK2: Participants with LRRK2-mutations but without Parkinson's symptoms
- no PD + no LRRK2: Participants without mutations and without Parkinson's symptoms
- PD+ other than LRRK2: Parkinson patients with mutations in other genes than LRRK2
- PD+ no LRRK2: Patients with idiopathic Parkinson's disease

SUMMARY:
The study aims to identify and systematically characterize Parkinson's patients with mutations in the LRRK2 gene. In about 90% of Parkinson's patients the cause of the disease is unclear. Based on current knowledge, it can be assumed that there are several causes and that the causes may be differ between patients; this makes research into the pathogenesis and possible therapies very difficult. In the case of monogenic Parkinson's diseases, which are due to changes in one gene (e.g. LRRK2), the function of the gene and possible disease mechanisms can be investigated. LRRK2-associated Parkinson's syndrome is clinically indistinguishable from idiopathic Parkinson's disease. It is inherited autosomal dominant, that means if one of the two gene copies is altered, the disease occurs. However, the disease does not occur in every mutation carrier, the penetrance is reduced and the mechanisms for that are still unclear. Ideally, knowledge of what influences penetrance could make it possible to exert targeted influence and prevent the disease. The comprehensive investigation of mechanisms of reduced penetrance but also of the effects of the mutation itself requires systematic investigations of as many affected persons as possible. We therefore aim to identify 4,000 people internationally, of them 1,500 with LRRK2-associated Parkinson's syndrome, 500 with LRRK2-mutations but without Parkinson's symptoms, 500 without mutations and without Parkinson's symptoms, 500 Parkinson patients with mutations in other genes than LRRK2 and 1,000 patients with idiopathic Parkinson's disease from the same populations. The participants will undergo a comprehensive survey on Parkinson's symptoms, concomitant diseases, environmental factors and medication and there is the possibility of more detailed genetic examinations. Participants will be asked to donate samples of blood, urine and household dust.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant.
* The participant is clinically diagnosed with Parkinson's disease or the individual is a family member of a participant with LRRK2 parkinsonism or is a member of a high risk population with an early PD onset.
* The participant is equal to or older than 18 years old.

Exclusion Criteria:

* Inability to provide informed consent.
* The participant is not suffering from Parkinson's disease or the individual is not a family member of a participant with LRRK2 parkinsonism or is not a member of a high risk population.
* The participant is younger than 18 years old.
* Previously enrolled in the study.
* Participant in custody.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease or family members of participants with LRRK2 parkinsonism or members of a high risk population with an early PD onset, able to provide informed consent and equal or older than 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiology of LRRK2-positive patients | 2 years
  Description of the frequency of all important clinical signs and symptoms including non-motor signs and factoring in the most important influencing factors such as sex, disease duration, and medication. We will report raw and corrected frequencies with 95% confidence intervals.

SECONDARY OUTCOMES:
Analysis of penetrance of LRRK2 mutations | 2 years
  Penetrance rates (the proportion of individuals with LRRL2 mutation who exhibit clinical symptoms of Parkinson's disease) and phenotypes, and will try to predict penetrance in logistic regression models and quantify the influence of different factors impacting on penetrance.
Analysis of expressivity of LRRK2 mutations | 2 years
  We will analyze expressivity (the degree in which a genotype is phenotypically expressed) of LRRK2 mutations. We will first define meaningful categories using our phenotypic data and then proceed to identify influencing factors.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Klein, Prof. Dr., Principal Investigator — Institute of Neurogenetics, University of Luebeck; Meike Kasten, Prof. Dr., Principal Investigator — Department of Psychiatry, University of Luebeck
Locations (1):
- Institute of Neurogenetics, Lübeck, Schelswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No
The Plan will be defined at later stages.

REFERENCES:
- [Derived] Usnich T, Vollstedt EJ, Schell N, Skrahina V, Bogdanovic X, Gaber H, Forster TM, Heuer A, Koleva-Alazeh N, Csoti I, Basak AN, Ertan S, Genc G, Bauer P, Lohmann K, Grunewald A, Schymanski EL, Trinh J, Schaake S, Berg D, Gruber D, Isaacson SH, Kuhn AA, Mollenhauer B, Pedrosa DJ, Reetz K, Sammler EM, Valente EM, Valzania F, Volkmann J, Zittel S, Bruggemann N, Kasten M, Rolfs A, Klein C; LIPAD Study Group. LIPAD (LRRK2/Luebeck International Parkinson's Disease) Study Protocol: Deep Phenotyping of an International Genetic Cohort. Front Neurol. 2021 Aug 9;12:710572. doi: 10.3389/fneur.2021.710572. eCollection 2021. PMID 34475849